CLINICAL TRIAL: NCT01280136
Title: Web-Based Middle School HIV Prevention Curricula: Aspiring for Reach and Impact
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Melissa Peskin, Assitant Professor - Health Promotion & Behavioral Science, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R01MH085594 (NIH); R01MH085594 (NIH)
Record Dates: First submitted 2011-01-14; First posted 2011-01-20 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: HIV; Sexually Transmitted Diseases
Keywords: HIV; Sexually Transmitted Diseases; Pregnancy Prevention; Abstinence Education; Adolescents; Sexual Health
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- It's Your Game Tech (Experimental): An interactive web-based HIV, sexually transmitted infection (STI), and pregnancy prevention program for 8th grade students. This web-based intervention will be adapted from the computer-based component of an existing successful prevention program, It's Your Game…Keep it Real, (IYG) as well as include critical elements from the IYG classroom component. The web-based intervention will consist of 13 lessons and will tailor information to the individual's gender and to his/her intentions or behaviors related to sexual risk-taking. The program will address peer norms, attitudes, self-efficacy, refusal skills, and communication skills related to healthy relationships, dating, and sexual risk-taking behavior.
  Interventions: Behavioral: It's Your Game Tech

INTERVENTIONS:
Behavioral: It's Your Game Tech — An interactive web-based intervention for 8th grade students. This web-based intervention will be adapted from the computer-based component of an existing successful prevention program, It's Your Game…Keep it Real, (IYG) as well as include critical elements from the IYG classroom component. The web-based intervention will consist of 13 lessons and will tailor information to the individual's gender and to his/her intentions or behaviors related to sexual risk-taking. The program will address peer norms, attitudes, self-efficacy, refusal skills, and communication skills related to healthy relationships, dating, and sexual risk-taking behavior.
  Other Names: IYG Tech

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a web-based HIV, sexually transmitted infection (STI), and pregnancy prevention curriculum as a stand alone intervention for 8th grade students in a large urban school district. This web-based curriculum will be adapted from the computer-based component of an existing successful prevention program, It's Your Game…Keep it Real, (IYG) but will be enhanced to include critical elements from the IYG classroom component. The primary hypothesis to be tested is: (1) students who receive the web-based curriculum will delay sexual activity relative to those who receive standard care. The major dependent variable is the proportion of students initiating sexual activity (vaginal, oral, or anal sex). Secondary hypotheses will examine the effect of the web-based curriculum on specific types of sex (e.g., vaginal, oral, anal) and psychosocial variables such as students' intentions, knowledge, self-efficacy, attitudes, and perceived norms related to sexual risk-taking behavior. Secondary hypotheses will also examine the effect of the intervention on the proportion of students who are sexually active, number of times students engage in unprotected sexual intercourse, and students' number of sexual partners.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of a web-based HIV, sexually transmitted infection (STI), and pregnancy prevention curriculum as a stand alone intervention for 8th grade students in a large urban school district. Twenty middle schools were invited to participate in the study. From those schools, we randomized 10 to the intervention group and 10 to the comparison condition, and will then recruit a cohort of 2,000 8th grade students into the study. Parental permission and youth assent will be required prior to participation. Students will be asked to complete a baseline and 12-month follow-up survey. The web-based curriculum will be adapted from the computer-based component of an existing successful prevention program, It's Your Game…Keep it Real, (IYG) but will be enhanced to include critical elements from the IYG classroom component. The web-based intervention will consist of 13 lessons and will tailor information to the individual's gender and to his/her intentions or behaviors related to sexual risk-taking. The program will address peer norms, attitudes, self-efficacy, refusal skills, and communication skills related to healthy relationships, dating, and sexual risk-taking behavior. The primary hypothesis to be tested is: (1) students who receive the web-based curriculum will delay sexual activity relative to those who receive standard care. The major dependent variable is the proportion of students initiating sexual activity (vaginal, oral, or anal sex). Secondary hypotheses will examine the effect of the web-based curriculum on specific types of sex (e.g., vaginal, oral, anal) and psychosocial variables such as students' intentions, knowledge, self-efficacy, attitudes, and perceived norms related to sexual risk-taking behavior. Secondary hypotheses will also examine the effect of the intervention on the proportion of students who are sexually active, number of times students engage in unprotected sexual intercourse, and students' number of sexual partners.

ELIGIBILITY:
Inclusion Criteria:

* 8th graders attending regular classes in large urban school district in Southeast Texas

Exclusion Criteria:

* No students will be excluded based on race/ethnicity, age, or gender
* Students will be informed that the surveys and intervention will only be available in English and will be asked to consider their comfort level with participating in the study.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1700 (Actual)
Dates: Start 2009-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
sexual initiation | baseline prior to intervention
sexual initiation | 12 month follow-up

SECONDARY OUTCOMES:
sexual activity in past 3 months | baseline prior to intervention
unprotected sexual intercourse | baseline prior to intervention
number of sexual partners | baseline prior to intervention
sexual activity in past 3 months | 12 month follow-up
unprotected sexual intercourse | 12 month follow-up
number of sexual partners | 12 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Peskin, PhD, Principal Investigator — University of Texas Houston School of Public Health; Ross Shegog, PhD, Principal Investigator — University of Texas Houston School of Public Health
Locations (1):
- University of Texas Houston School of Public Health, Houston, Texas, United States